CLINICAL TRIAL: NCT06344780
Title: A Multi-center Study of the Clinical Outcomes of Abemaciclib, Palbociclib or Dalpiciclib Combined with Endocrine Therapy As First-line Treatment in HR Positive, HER2 Negative Unresectable or Metastatic Breast Cancer in Real World Practice
Brief Title: Abemaciclib, Palbociclib or Dalpiciclib Combined with Endocrine Therapy As First-line Treatment in HR Positive, HER2 Negative Unresectable or Metastatic Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-28
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Abemaciclib; Palbociclib; Dalpiciclib; HR Positive; HER2 Negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Abemaciclib cohort
- Palbociclib cohort
- Dalpiciclib cohort

SUMMARY:
A multi-center, real world study to evaluate the clinical outcomes and safety of Abemaciclib, Palbociclib or Dalpiciclib combined with endocrine therapy as first-line treatment in HR Positive, HER2 Negative unresectable or metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 18 years old;
2. Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between June 2020 to October 2023;
3. Received CDK4/6 inhibitors(Abemaciclib, Palbociclib or Dalpiciclib) as first-line therapy for at least one cycle;
4. Complete medical history was available.

Exclusion Criteria:

1. Medical history was incomplete.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between June 2020 to October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Pregression-free survival

SECONDARY OUTCOMES:
OS | 6 weeks
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen Y, Xie Y, Sang D, Xie N, Han X, Zhao Y, Li J, Yue J, Yuan P, Wang B. Real-world comparison of palbociclib, abemaciclib, and dalpiciclib as first-line treatments for Chinese HR+/HER2-metastatic breast cancer patients: a multicenter study (YOUNGBC-28). Ther Adv Med Oncol. 2024 Dec 17;16:17588359241302018. doi: 10.1177/17588359241302018. eCollection 2024. PMID 39697620